CLINICAL TRIAL: NCT03582722
Title: Use of a Weight Loss Aid in a Population Exposed to Polybrominated Biphenyls (PBB)
Brief Title: Weight Loss Aid in an Exposed Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Healthway Compounding Pharmacy (Industry); Michigan Public Health Departments (Other Government); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Michele Marcus, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00099231; R01ES025775 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: Polybrominated Biphenyl Poisoning
Keywords: Polybrominated Biphenyl Exposure; Gastrointestinal lipase inhibitor
MeSH Terms: interventions — Orlistat; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orlistat Weight Loss Aid (Experimental): Participants randomized to take orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin will also be recommended and monitored.
  Interventions: Drug: Orlistat; Dietary Supplement: Multivitamin
- Placebo (Placebo Comparator): Participants randomized to take a placebo to match orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin will also be recommended and monitored.
  Interventions: Drug: Placebo capsule; Dietary Supplement: Multivitamin

INTERVENTIONS:
Drug: Orlistat — Participants will be instructed to take one 60mg capsule of orlistat with each meal containing fat, up to three capsules daily, for six months.
  Other Names: Alli
  Arms: Orlistat Weight Loss Aid
Drug: Placebo capsule — Participants will be instructed to take one placebo capsule to match 60mg of orlistat with each meal containing fat, up to three capsules daily, for six months.
  Arms: Placebo
Dietary Supplement: Multivitamin — A multivitamin will be provided to be taken once daily, at bedtime.

SUMMARY:
This study will explore whether the use of orlistat results in weight loss that is accompanied by a reduction in the body burdens of polybrominated biphenyls (PBB) and other Persistent Organic Pollutants (POPs).

DETAILED DESCRIPTION:
Millions of people living in Michigan were exposed to brominated flame retardants (polybrominated biphenyls or PBB) as a result of the largest agricultural disaster in US history. Over the past six years, Emory researchers have tested nearly 900 Michigan residents and determined that 60% still had PBB in their bodies from that disaster. PBB is stored in body fat and the researchers at Emory have been asked by community members if weight loss might reduce their body burdens of PBB and other lipophilic chemicals. In an effort to understand how PBB and other persistent organic pollutants (POPs) are eliminated, the researchers are conducting a randomized trial of orlistat versus placebo.

Orlistat is an over-the-counter product approved by the FDA for weight loss and works by increasing excretion of fat into the stool. Since PBB is stored in body fat, the researchers hypothesize that orlistat may reduce the body burden of PBB and other POPs. This study is a randomized, placebo-controlled trial of orlistat (at the dose available over-the-counter) plus diet and exercise for 6 months in a population with elevated PBB levels. Participants will be healthy overweight adults and orlistat will be taken as directed for the approved indication (weight loss).

ELIGIBILITY:
Inclusion Criteria:

* current or recent (within the last five years) serum PBB level of ≥1ppb, or are a member of a sub-group likely to have high serum PBB (former chemical worker, family member of former chemical worker, lived on a farm with animals that were quarantined because of PBB exposure)
* at least 18 years old
* currently reside in Michigan
* able to participate in examinations and laboratory tests (a lipid panel, liver function test, thyroid function and and creatinine levels) done at at a local health department or other medical health facility and to be able to engage in moderate physical activity (e.g. walking)
* participants with undiagnosed abdominal pain or diarrhea, Crohn's disease, Ulcerative Colitis, Celiac Disease, treated diabetes or treated thyroid disorder, will only be eligible following consultation with their primary care provider
* any participant using levothyroxine will be instructed to take their dosage 4 hours before or after Orlistat in order to maintain eligibility

Exclusion Criteria:

* BMI<25
* abnormal liver function
* abnormal creatinine levels
* abnormal thyroid levels (TSH)
* have type 1 diabetes
* have had an organ transplant
* are pregnant or lactating
* current use of weight-loss medications, oral steroids, Coumadin, warfarin or Cyclosporine
* have a diagnosed problem absorbing food, or have an eating disorder
* a history of bariatric surgery, pancreatitis, kidney stones, gall bladder disorder or a serious chronic disease (e.g. uncontrolled diabetes, congestive heart failure, chronic kidney disease)
* allergies to any ingredients of the Orlistat over-the-counter (OTC) capsules
* participants will become ineligible at any point during the study if they begin a medical regimen involving any of the above medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Marcus, PhD, MPH, Principal Investigator — School of Public Health, Emory University
Locations (1):
- Michele Marcus, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Michigan polybrominated biphenyls (PBB) Research Registry. Participant enrollment began September 14, 2018 and all follow-up assessments were completed by June 30, 2022.
Pre-assignment Details: 100 individuals gave consent to participate in the study and were randomized to a study arm. One participant who was randomized to the Orlistat arm did not begin taking the study medication and did not complete the first study visit.
Groups:
- Placebo: Participants randomized to take a placebo to match orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin were also recommended and monitored.
  Placebo capsule: Participants were instructed to take one placebo capsule to match 60mg of orlistat with each meal containing fat, up to three capsules daily, for six months.
  Multivitamin: A multivitamin was provided to be taken once daily, at bedtime.
- Orlistat Weight Loss Aid: Participants randomized to take orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin were also recommended and monitored.
  Orlistat: Participants were instructed to take one 60mg capsule of orlistat with each meal containing fat, up to three capsules daily, for six months.
  Multivitamin: A multivitamin was provided to be taken once daily, at bedtime.
Period: Overall Study
Arm/Group | Placebo | Orlistat Weight Loss Aid
Started (Individuals who gave consent to participate and were randomized to a study arm.) | 49 | 51
Completed the Enrollment Visit and Initiated Study Medication | 49 | 50
Completed the 3 Month Follow-up Visit (Participants who completed at least a 3-month follow-up visit are included in the outcome tables (n=91).) | 46 | 45
Completed (Completed the 6 month follow-up visit. Two people who completed the 3-month visit but not the 6-month visit are included in the outcome tables.) | 45 | 44
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes participants who completed both the Enrollment visit and the Month 3 visit.
Groups:
- Placebo: Participants randomized to take a placebo to match orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin were also recommended and monitored.
- Orlistat Weight Loss Aid: Participants randomized to take orlistat at the over-the-counter dose for six months. Diet and exercise plus a daily multivitamin were also recommended and monitored.
- Total: Total of all reporting groups
Arm/Group | Placebo | Orlistat Weight Loss Aid | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.9) | 59.5 (9.3) | 59.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 46 | 43 | 89
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 43 | 86
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Participant weight, in kilograms, was measured in light clothing without shoes on a regularly calibrated digital scale.
Time Frame: Enrollment, Month 3, Month 6
Population: This analysis includes participants who attended both the Enrollment and Month 3 visits, and also those who completed the Month 6 visit. Twenty-five participants were not able to attend the Month 3 study visit in person; 23 due to the Coronavirus 2019 (COVID-19) pandemic and an additional 2 due to other reasons. All of participants who were unable to have the in-person Month 3 visit provided a self-measured weight. Mean weights measured per protocol and self-measured are reported separately.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
kilograms (kg)
  Enrollment | 91.3 (16.4) | 92.3 (17.8)
  Month 3 measured per protocol by study staff: number analyzed (Participants) | 33 | 33
  Month 3 measured per protocol by study staff | 88.6 (18.1) | 87.4 (15.9)
  Month 3 self-measured by participant: number analyzed (Participants) | 13 | 12
  Month 3 self-measured by participant | 90.4 (14.1) | 93.2 (20.2)
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 89.2 (17.1) | 88.1 (17.7)

2. Primary Outcome: Body Mass Index (BMI)
Description: Body Mass Index is a weight-to-height ratio, calculated by dividing one's weight in kilograms by the square of one's height in meters and used as an indicator of obesity and underweight. Participants had their weight measured in light clothing without shoes on a regularly calibrated digital scale. Height is measured using a well-mounted stadiometer.
Time Frame: Enrollment, Month 3, Month 6
Population: This analysis includes participants who attended both the Enrollment and Month 3 visits, and also those who completed the Month 6 visit. Twenty-five participants were not able to attend the Month 3 study visit in person; 23 due to the COVID-19 pandemic and an additional 2 due to other reasons. All of participants who were unable to have the in-person Month 3 visit provided a self-measured weight. Mean BMI calculated using weight measured per protocol and self-measured are reported separately.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
kg/m^2
  Enrollment | 32.3 (5.4) | 31.7 (5.0)
  Month 3 - BMI calculated with weight measured by study staff: number analyzed (Participants) | 33 | 33
  Month 3 - BMI calculated with weight measured by study staff | 31.5 (5.9) | 29.9 (4.1)
  Month 3 - BMI calculated with weight self-measured by participant: number analyzed (Participants) | 13 | 12
  Month 3 - BMI calculated with weight self-measured by participant | 31.6 (5.6) | 32.3 (6.4)
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 31.4 (5.8) | 30.2 (5.0)

3. Secondary Outcome: Serum Concentration of Polybrominated Biphenyl (PBB) 153
Description: PBB is an organic bromine compound that is environmentally toxic and is classified as a persistent organic pollutant. PBB 153 concentration in serum is measured in nanograms per milliliter (ng/mL).
Time Frame: Enrollment, Month 3, Month 6
Population: This analysis includes participants who attended both the Enrollment and Month 3 visits, and also those who completed the Month 6 visit. Twenty-three participants were not able to attend the Month 3 study visit in person due to the COVID-19 pandemic and did not have blood drawn at this time point. An additional 2 participants did not attend the Month 3 visit in person and one had blood collected and shipped to the study lab by their physician.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.454 [0.156 to 1.711] | 0.276 [0.145 to 0.751]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.355 [0.084 to 1.846] | 0.395 [0.201 to 0.801]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.481 [0.121 to 1.510] | 0.290 [0.131 to 0.889]

4. Secondary Outcome: Serum Concentration of Polybrominated Diphenyl Ether (PBDE) 47
Description: PBDE is an organic bromine compound that is environmentally toxic and is classified as a persistent organic pollutant. PBDE 47 concentration in serum is measured in ng/mL.
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.032 [0.015 to 0.059] | 0.028 [0.016 to 0.053]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.034 [0.015 to 0.057] | 0.025 [0.009 to 0.047]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.029 [0.017 to 0.056] | 0.025 [0.012 to 0.047]

5. Secondary Outcome: Serum Concentration of Polychlorinated Biphenyl (PCB) 118
Description: PCB is an organic chlorine compound that is environmentally toxic and is classified as a persistent organic pollutant. PCB 118 concentration in serum is measured in ng/mL.
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.035 [0.021 to 0.056] | 0.026 [0.014 to 0.041]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.031 [0.014 to 0.049] | 0.024 [0.014 to 0.044]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.028 [0.020 to 0.042] | 0.025 [0.014 to 0.044]

6. Secondary Outcome: Serum Concentration of PCB 138
Description: PCB is an organic chlorine compound that is environmentally toxic and is classified as a persistent organic pollutant. PCB 138 concentration in serum is measured in ng/mL
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.081 [0.039 to 0.119] | 0.064 [0.040 to 0.111]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.070 [0.030 to 0.109] | 0.066 [0.039 to 0.120]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.078 [0.036 to 0.108] | 0.064 [0.042 to 0.129]

7. Secondary Outcome: Serum Concentration of PCB 153
Description: PCB is an organic chlorine compound that is environmentally toxic and is classified as a persistent organic pollutant. PCB 153 concentration in serum is measured in ng/mL.
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.122 [0.060 to 0.184] | 0.096 [0.062 to 0.166]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.100 [0.039 to 0.185] | 0.105 [0.059 to 0.179]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.114 [0.061 to 0.191] | 0.105 [0.064 to 0.178]

8. Secondary Outcome: Serum Concentration of PCB 180
Description: PCB is an organic chlorine compound that is environmentally toxic and is classified as a persistent organic pollutant. PCB 180 concentration in serum is measured in ng/mL
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.116 [0.064 to 0.188] | 0.108 [0.076 to 0.165]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.101 [0.050 to 0.214] | 0.114 [0.074 to 0.177]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.112 [0.060 to 0.190] | 0.121 [0.071 to 0.187]

9. Secondary Outcome: Serum Concentration of Dichlorodiphenyldichloroethylene (DDE)
Description: DDE is a chemical produced by the breakdown of dichlorodiphenyltrichloroethane (DDT). High levels of DDE can impact lactation and increase the risk of preterm birth. DDE concentration in serum is measured in ng/mL.
Time Frame: Enrollment, Month 3, Month 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Orlistat Weight Loss Aid
Number analyzed (Participants) | 46 | 45
ng/mL
  Enrollment | 0.535 [0.343 to 0.844] | 0.490 [0.336 to 0.686]
  Month 3: number analyzed (Participants) | 33 | 34
  Month 3 | 0.539 [0.305 to 1.005] | 0.490 [0.360 to 0.735]
  Month 6: number analyzed (Participants) | 45 | 44
  Month 6 | 0.573 [0.318 to 0.874] | 0.498 [0.359 to 0.768]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time individuals gave consent to participate in the study and continued through the 6 Month study visit.
Arm/Group | Placebo | Orlistat Weight Loss Aid
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 3/49 | 0/51
Other Adverse Events (participants affected / at risk) | 28/49 | 41/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | Orlistat Weight Loss Aid (N=51)
Heart attack (Cardiac disorders) | 1 | 0
Hospitalization due to allergic reaction to an antibiotic (General disorders) | 1 | 0
Abdominal pain; masses on ovary, liver, and kidney; endometriosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | Orlistat Weight Loss Aid (N=51)
Headache (General disorders) | 5 | 6
Dizziness (General disorders) | 0 | 3
Diarrhea and frequent or oily bowel movements (Gastrointestinal disorders) | 13 | 28
Stomach ache or gassy (Gastrointestinal disorders) | 5 | 1
Cold/flu/respiratory symptoms (Infections and infestations) | 12 | 14
COVID-19 (Infections and infestations) | 3 | 2
Falls (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03582722/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03582722/ICF_000.pdf